CLINICAL TRIAL: NCT05138926
Title: Immediate Effect of High Speed and Low Amplitude Cervical Manipulation on the Electromyographic Activity of the Masseter Muscle, in a Physiotherapy Students at the University of the Americas. a Clinical Trial, Single Blind
Brief Title: Effect of Spinal Manipulation on Electromyography of the Masseter Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Americas (Other)
Responsible Party: Principal Investigator, Ignacio Astudillo Ganora, Physiotherapist, Phd, University of Americas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEC_FP_2021027
Record Dates: First submitted 2021-11-16; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Bruxism; Muscle Disorder
MeSH Terms: conditions — Bruxism; Muscular Diseases | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical manipulation group (Experimental): high speed, low amplitude cervical manipulation
  Interventions: Other: Cervical Manipulation
- Control group (Sham Comparator): placebo mobilization without manipulation
  Interventions: Other: Sham Cervical Manipulation

INTERVENTIONS:
Other: Cervical Manipulation — high speed, low amplitude cervical manipulation
  Arms: Cervical manipulation group
Other: Sham Cervical Manipulation — Cervical mobilization without performing spinal manipulation
  Arms: Control group

SUMMARY:
Research Problem: To know the immediate effects of high speed and low amplitude cervical manipulation on the electromyographic activity of the masseter muscles of physiotherapy students at the University of the Americas Course objective: To compare the immediate effects of high-speed, low-amplitude cervical manipulation on the electromyographic activity of the masseter muscles versus a placebo intervention in kinesiology students at the University of the Americas.

Specific objectives: To describe the changes in the electromyographic activity of the masseter muscles of the high-speed cervical manipulation group in students of the physiotherapy school of the University of the Americas of the Santiago Centro campus.

To describe the changes in the electromyographic activity of the masseter muscles of the placebo group in students of the physiotherapy school of the University of the Americas of the Santiago Centro campus.

Methodology: Single-blind, randomized clinical trial. Expected results: Significant differences are expected between the intervention group and the control group. This is reflected in a decrease in electromyographic activity in the masseter muscles after high-speed cervical manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female physiotherapy students over 18 years of age who regularly attend face-to-face classes who have a mobility pass and a health declaration.
* Students who read and sign the informed consent.

Exclusion Criteria:

* Orthognathic surgery.

  * Recent head and neck injury or fracture (equal to or less than 3 months)
  * Dental or medical diagnosis of mandibular disorder or manifest facial pain.
  * Contraindication (red flag) to perform high speed and low amplitude cervical manipulation (bone cancer, osteoporosis, vertebral artery injury, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Electromyography of the masseter muscle before intervention | baseline
  surface electromyography of the masseter muscle, measured in millivolts (mV)
Electromyography of the masseter muscle after the intervention | 5 minute after intervention
  surface electromyography of the masseter muscle, measured in millivolts (mV)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de las Americas, Santiago, Santiago Metropolitan, Chile